CLINICAL TRIAL: NCT02635360
Title: A Randomized Phase II Study of Chemoradiation and Pembrolizumab for Locally Advanced Cancer
Brief Title: Pembrolizumab and Chemoradiation Treatment for Advanced Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Linda R Duska (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Linda R Duska, Associate Professor, Division of Gynecology Oncology, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18472; UVA-LACC-PD201 (Other Grant/Funding Number: Merck Sharp & Dohme Corp.)
Record Dates: First submitted 2015-12-04; First posted 2015-12-18 (Estimated); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Cervical Cancer
Keywords: advanced; cervical cancer; pembrolizumab; chemoradiation; immunotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — pembrolizumab; Brachytherapy; Chemoradiotherapy; Cisplatin; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Following chemoradiation (Experimental): Subjects will receive standard chemotherapy weekly and 4-6 fractions of brachytherapy radiation for 5-6 weeks. After chemoradiation is complete, subjects will receive the study drug, pembrolizumab.
  Interventions: Drug: Pembrolizumab; Radiation: Brachytherapy; Drug: Cisplatin
- Concurrent to chemoradiation (Experimental): Subjects will receive standard chemotherapy weekly and 4-6 fractions of brachytherapy radiation for 5-6 weeks. While subjects are receiving chemotherapy and radiation, they will also receive the study drug, pembrolizumab.
  Interventions: Drug: Pembrolizumab; Radiation: Brachytherapy; Drug: Cisplatin

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg of study drug is given through intravenous (IV) administration once every 21 days for 3 months.
  Other Names: Keytruda; MK-3475
Radiation: Brachytherapy — Radiation is done for standard clinical care purposes.
  Other Names: chemoradiation
Drug: Cisplatin — 40 mg of chemotherapy drug will be given weekly for 5-6 weeks.
  Other Names: chemotherapy

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of immunotherapy in combination with chemotherapy and radiation (chemoradiation) for the treatment of advanced cervical cancer. Pembrolizumab, a type of immunotherapy called a checkpoint inhibitor, will be administered after or during chemoradiation.

DETAILED DESCRIPTION:
Primary: (1) To estimate the immunologic effects, as assessed in the tumor & PBMC, of both sequential and concurrent administration of pembrolizumab to CRT. Change between pre and post measurements of HPV E2, E7 specific CD8+ T cells, regulatory FoxP3+ T cells (Tregs) and the ratio of CD8+ T cells to Tregs are the immune measurements of primary interest. (2) To determine the safety of concurrent chemoradiation in combination with pembrolizumab for the treatment of locally advanced cervical cancer. Secondary: (1) To estimate rates of complete metabolic response on PET/CT imaging obtained 12 weeks after CRT.

(2) To estimate rates of distant metastasis as the first site of recurrence for patients.

(3) To estimate the influence of concurrent and consolidative MK-3475 on levels of plasminogen activator inhibitor-1 (PAI-1), a marker of immunosuppressive TGF-B.

(4) To estimate the influence of concurrent and consolidative MK-3475 on levels of IDO, an enzyme that depletes tryptophan, which is essential for T-cell function.

(5) To estimate the influence of concurrent and consolidative MK-3475 on levels of MHC class I (CD8+ T cell ligand) and MICA (NK ligand), as measured by MHC.

(6) To estimate the progression free survival (PFS) in subjects with locally advanced cervical cancer treated with sequential and concurrent administration of pembrolizumab in relation to CRT.

(7) To estimate the overall survival (OS) in subjects with locally advanced cervical cancer treated with sequential and concurrent administration of pembrolizumab in relation to CRT.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed cervical cancer.
* Must have adequate organ function.

Exclusion Criteria:

* Subject is pregnant.
* Recurrent cervical cancer.
* Distant metastases.
* Malignancy within the last 5 years; basal cell carcinoma or squamous cell carcinoma of the skin that has undergone potentially curative therapy is permissable.
* Subject has had prior radiation, chemotherapy, targeted therapy, or investigational therapy for cervical cancer.
* Subject has a immunodeficiency.
* Known history of HIV, Hepatitis B, Hepatitis C, TB, or inflammatory bowel disease.
* Hypersensitivity to pembrolizumab or similar drugs.
* Subject has an active autoimmune disease in the past 2 years.
* Known history of non-infectious pneumonitis.
* Subject has an active infection.
* Subject has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases are permissible. Talk to Study Contact for specifics.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Duska, MD, Principal Investigator — University of Virginia
Locations (8):
- United States (8):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Johns Hopkins, Baltimore, Maryland
  - Washington University, School of Medicine, St Louis, Missouri
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Virginia, Charlottesville, Virginia
  - INOVA Fairfax Hospital, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Derived] Lin AJ, Dehdashti F, Massad LS, Thaker PH, Powell MA, Mutch DG, Schwarz JK, Markovina S, Siegel BA, Grigsby PW. Long-Term Outcomes of Cervical Cancer Patients Treated With Definitive Chemoradiation Following a Complete Metabolic Response. Clin Oncol (R Coll Radiol). 2021 May;33(5):300-306. doi: 10.1016/j.clon.2021.01.010. Epub 2021 Feb 11. PMID 33581976

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Following Chemoradiation | Concurrent to Chemoradiation
Started | 48 | 46
Completed | 42 | 39
Not Completed | 6 | 7
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Non-Compliance | 3 | 1
Not completed — Disease Progression | 0 | 2
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Following Chemoradiation | Concurrent to Chemoradiation | Total
Number analyzed (Participants) | 48 | 46 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 44 | 87
  >=65 years | 5 | 2 | 7
Age, Continuous [Mean (Full Range); unit: years] | 49 [29 to 77] | 48 [28 to 76] | 48 [28 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 46 | 94
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 42 | 38 | 80
  Unknown or Not Reported | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 9 | 6 | 15
  White | 28 | 37 | 65
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 48 | 46 | 94

OUTCOME MEASURES:

1. Primary Outcome: Change in Immunologic Markers Following Combination of Study Drug With Chemoradiation
Description: Expression of immune markers measured at pre and post administration of study drug with chemoradiation will be compared, analyzed and enumerated using QuPath software to provide a cell #/mm2 (not per high power field) and the ratio of CD8+ cells:FoxP3+ cells/mm2 was calculated.
Time Frame: 12 weeks post-chemoradiation
Measure: Mean (Standard Deviation); unit: ratio of cells per mm^2", "CD8+: FoxP3+
Arm/Group | Following Chemoradiation | Concurrent to Chemoradiation
Number analyzed (Participants) | 37 | 28
ratio of cells per mm^2", "CD8+: FoxP3+ | 31.31 (124.77) | 140.33 (812.53)

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: To determine the safety of concurrent chemoradiation in combination with pembrolizumab for the treatment of locally advanced cervical cancer
Time Frame: From start of treatment until 12 weeks post-chemoradiation
Population: Subjects on Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Following Chemoradiation | Concurrent to Chemoradiation
Number analyzed (Participants) | 48 | 46
Participants | 0 | 4

3. Secondary Outcome: Metabolic Response Rate on PET/CT Imaging
Description: To estimate rates of complete metabolic response on PET/CT imaging obtained 12 weeks after CRT
Time Frame: 12 weeks after chemotherapy
Population: Subjects that completed Radiation Therapy within 56 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Following Chemoradiation | Concurrent to Chemoradiation
Number analyzed (Participants) | 33 | 34
Participants | 2 | 7

4. Secondary Outcome: Incidence of Distant Metastases
Description: To estimate the rates of distant metastasis as the first site of recurrent for patients
Time Frame: From start of treatment until up to 5 years following end of treatment
Population: Number of subjects on treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Following Chemoradiation | Concurrent to Chemoradiation
Number analyzed (Participants) | 48 | 46
Participants | 6 | 6

5. Secondary Outcome: Progression Free Survival
Description: To estimate the progression free survival (PFS) in subjects with locally advanced cervical cancer treatment with sequential and concurrent administration of pembrolizumab in relation to CRT
Time Frame: From start of treatment until up to 5 years following end of treatment
Population: Number of Subjects on Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Following Chemoradiation | Concurrent to Chemoradiation
Number analyzed (Participants) | 48 | 46
Participants | 41 | 38

6. Secondary Outcome: Overall Survival
Description: To estimate the overall survival (OS) in subjects with locally advanced cervical cancer treated with sequential and concurrent administration of pembrolizumab in relation to CRT
Time Frame: From start of treatment until up to 5 years following end of treatment
Population: Number of subjects on treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Following Chemoradiation | Concurrent to Chemoradiation
Number analyzed (Participants) | 48 | 46
Participants | 42 | 41

ADVERSE EVENTS:
Time Frame: Start of treatment (week 1) through end of treatment visit (35 +/- 5 days following the final treatment).
Description: Adverse experiences will be graded according to NCI CTCAE Version 4.0. Toxicities will be characterized in terms regarding seriousness, causality, toxicity grading and action taken with regard to trial treatment. All adverse events will be reported according per protocol. Throughout the study, investigators should report any deaths, serious adverse events or other adverse events of concern they believe to be related to the investigational agent.
Arm/Group | Following Chemoradiation | Concurrent to Chemoradiation
All-Cause Mortality (participants affected / at risk) | 8/48 | 5/46
Serious Adverse Events (participants affected / at risk) | 40/48 | 27/46
Other Adverse Events (participants affected / at risk) | 18/48 | 11/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Following Chemoradiation (N=48) | Concurrent to Chemoradiation (N=46)
Anemia (Blood and lymphatic system disorders) | 2 | 5
Atrial fibrillation (Cardiac disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 2
Gastrointestinal Pain (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 8
Vomitng (Gastrointestinal disorders) | 3 | 4
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Allergic Reaction (Immune system disorders) | 1 | 0
Kidney Infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 0
Urinary Tract Infection (Infections and infestations) | 4 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 2 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Colonic stenosis (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Flu like symptoms (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Following Chemoradiation (N=48) | Concurrent to Chemoradiation (N=46)
Nausea (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Fever (General disorders) | 4 | 3
Blurred Vision (Eye disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3
Urinary Tract Infection (Renal and urinary disorders) | 2 | 0
Creatinine increased (Investigations) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT02635360/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT02635360/ICF_001.pdf